CLINICAL TRIAL: NCT03336983
Title: Bone Response After Luteinizing Hormone-releasing Hormone Analogue and Enzalutamide +/- Zoledronic Acid in Prostate Cancer Patients With Hormone Sensitive Metastatic Bone Disease: a Prospective, Phase II, Randomized, Multicenter Study
Brief Title: Luteinizing Hormone-releasing Hormone Analogue and Enzalutamide +/- Zoledronic Acid in Prostate Cancer Patients
Acronym: BonEnza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Alfredo Berruti, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCB-ONCO-2336-2017; 2017-000305-21 (EudraCT Number)
Record Dates: First submitted 2017-10-23; First posted 2017-11-08 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Bone Metastases
Keywords: prostate cancer; bone metastasis; enzalutamide; zoledronic acid
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid; enzalutamide

STUDY DESIGN:
Intervention Model Description: prostate cancer patients with hormone sensitive metastatic bone disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LHRH-A + Enzalutamide (Other): Prostate cancer patients with hormone sensitive metastatic bone disease will be treated with LHRH-A + Enzalutamide until patient's progression, consent withdrawal or unacceptable toxicity
  Interventions: Drug: Enzalutamide
- LHRH-A + Enzalutamide + Zoledronic Acid (Experimental): Prostate cancer patients with hormone sensitive metastatic bone disease will be treated with LHRH-A + Enzalutamide + Zoledronic Acid until patient's progression, consent withdrawal or unacceptable toxicity
  Interventions: Drug: Zoledronic Acid; Drug: Enzalutamide

INTERVENTIONS:
Drug: Zoledronic Acid — Prostate cancer patients with hormone sensitive metastatic bone disease will be treated with LHRH-A + Enzalutamide in the presence or absence of Zoledronic Acid
  Other Names: Zoledronate
  Arms: LHRH-A + Enzalutamide + Zoledronic Acid
Drug: Enzalutamide — Patients from both arms will be treated with LHRH-A + Enzalutamide
  Other Names: Xtandi

SUMMARY:
This study was undertaken to evaluate bone response in metastatic prostate cancer patients treated with Enzalutamide with or without Zoledronic Acid in combination with luteinizing hormone-releasing hormone (LHRH) analogue with the use of Whole Boby (WB) DW-MRI.

DETAILED DESCRIPTION:
Most men with fatal prostate cancer develop bone metastases and bone is often the dominant or the only site of metastatic disease. Bone metastases are an important cause of morbidity since they are associated with skeletal related events (SREs) including pathologic fractures, spinal cord compression, and need for surgery or radiation therapy to bone. Osteoclast-mediated bone destruction is the key pathologic mechanism for SREs in prostate cancer and other malignancies. Zoledronic acid (ZA) is a potent inhibitors of osteoclast-mediated bone resorption. ZA has demonstrated to be effective in preventing SREs in patients with castrate resistant disease; however, its efficacy in hormone naïve disease is uncertain.

In the last few years new drugs targeting directly the androgen receptor such as Enzalutamide have shown to be very effective in terms of survival prolongation in the management of castration resistant disease and the efficacy in hormone naïve patients is currently under investigation. Interestingly, the results of a large scale, prospective, randomized clinical trial have shown that Enzalutamide administration is also associated with a reduction in the risk of SREs and this raises the question of the usefulness of the addition of bone resorption inhibitors to Enzalutamide.

The evaluation of bone response of antineoplastic therapies has always been difficult in metastatic bone prostate cancer patients due to their osteoblastic nature. Whole body diffusion-weighted (DW) MRI has been recently proposed as new imaging tool for grading treatment response in patients with skeletal metastases from prostate cancer. According to the literature data DW images can allow the identification of bone marrow infiltration and tumor necrosis induced by treatment. In addition, this technique allows to monitor the bone marrow restoration. This, this technique was selected to evaluate bone response in metastatic prostate cancer patients treated with Enzalutamide with or without Zoledronic Acid in combination with LHRH-A.

Moreover, since androgen-receptor isoform encoded by splice variant 7 (AR-V7) is an androgens' receptor variant that could have a potential clinical utility as a prognostic factor and predictive marker of therapy response, an ancillary study will be conducted to evaluate ARV7 expression in Circulating Tumor Cells (CTC).

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of prostate carcinoma,
2. Age > 18 years,
3. Metastatic disease documented as the presence of bone lesions on bone scan associated or not to soft tissue lesions measurable at computed tomography (CT) scan or Magnetic Resonance Imaging (MRI),
4. No previous hormone or chemotherapeutic treatments given for prostate carcinoma (patients that are receiving LHRH-A therapy for less than 4 months are admitted),
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1,
6. Expected life expectancy ≥ 6 months,
7. Subject capable to swallow the Study's medication and to comply with the Study's requirements,
8. Signed informed consent.

Exclusion Criteria:

1. Presence of active serious disease, active infection or co-comorbidity that may prevent the study enrollment make (at the discretion of the clinical Investigator),
2. Known or suspected brain metastases or active leptomeningeal dissemination,
3. History of other malignant neoplasm during the previous 5 years, different from the non-melanoma skin carcinoma,
4. Absolute Neutrophil Count (ANC) < 1.500/µL, platelet < 100.000/µL, or hemoglobin < 5,6 mmol/L (< 9 g/dL) at Screening Visit (notably: patients must not receive neither any growth factor during the previous 7 days nor any blood transfusion during the 28 days preceding the hematology sampling performed at Screening),
5. Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2,5 x upper limit of normal (ULN) at Screening Visit,
6. Creatinine > 177 µmol/L (> 2 mg/dL) at Screening Visit,
7. Albumin ≤ 30 g/L (≤ 3,0 g/dL) at Screening Visit,
8. History of seizures or any other seizure-predisposed pathology; history of loss of consciousness or transitory ischaemic attack during the 12 months preceding the Screening visit,
9. Clinically significant cardiovascular disease including:

   * myocardial infarction (6 months preceding the screening)
   * uncontrolled angina (3 months preceding the screening)
   * Congestive heart failure New York Heart Association (NYHA) class 3 or 4, congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan performed within three months results in a left ventricular ejection fraction that is ≥ 45%;
   * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes);
   * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
   * Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mmHg) at the Screening visit;
   * Bradycardia as indicated by a heart rate of < 50 beats per minute on the Screening ECG;
   * Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the Screening visit;
10. Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months);
11. Major surgery within 4 weeks of enrollment (Day 1 Visit);
12. Radiation therapy for treatment of the primary tumor within 3 weeks of enrollment (Day 1 visit);
13. Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease Prostate-specific antigen (PSA) levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within four weeks of enrollment (Day 1 visit);
14. Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 126 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in bone response after 6 and 12 months of treatment compared to baseline | Exam will be performed at baseline and after 6 and 12 months of treatment
  Whole-body Diffusion MRI

SECONDARY OUTCOMES:
Evaluation of bone repair | Screening visit; 12 months of treatment
  CT Scan
Changes in bone mineral density after 18 months of treatment compared to baseline | Screening visit; 18 months of treatment
  Dual energy x-ray absorptiometry (DEXA Scan)
Functional Assessment of Cancer Therapy-Prostate | Monthly until end of treatment (18 months)
  Functional Assessment of Cancer Therapy-Prostate (FACT- P) Questionnaire will be collected from patients.It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain, as well as a global Qquality of Life (QoL) score.
Brief Pain Inventory-Short Form Questionnaire | Monthly until end of treatment (18 months)
  Brief Pain Inventory-Short Form (BPI-SF) Questionnaire will be collected from patients.In particular, a 0-10 numerical rating scale was used to measure pain severity items where 0=no pain and 10=pain as bad as you can imagine or with 0=pain did not interfere with my normal life and 10=pain interferes ompletely. A question about the percentage and duration of pain relief was also included.
Weight evaluation | Screening visit; 18 months of treatment
  Evaluation of patient weight expressed in kg after 18 months of treatment compared to baseline
C-terminal telopeptide analysis | Screening visit; 2, 4, 6, 9, 12, 18 months of treatment
  C-terminal telopeptide analysis (CTX, ng/ml) evaluation on peripheral blood samples
Bone alkaline phosphatase analysis | Screening visit; 2, 4, 6, 9, 12, 18 months of treatment
  Bone alkaline phosphatase analysis (U/uL) evaluation on peripheral blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, MD, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Azienda Ospedaliera Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt GP, Reiser MF, Baur-Melnyk A. Whole-body MRI for the staging and follow-up of patients with metastasis. Eur J Radiol. 2009 Jun;70(3):393-400. doi: 10.1016/j.ejrad.2009.03.045. Epub 2009 May 19. PMID 19457631
- [Background] Koh DM, Blackledge M, Padhani AR, Takahara T, Kwee TC, Leach MO, Collins DJ. Whole-body diffusion-weighted MRI: tips, tricks, and pitfalls. AJR Am J Roentgenol. 2012 Aug;199(2):252-62. doi: 10.2214/AJR.11.7866. PMID 22826385
- [Result] Smith MR, Halabi S, Ryan CJ, Hussain A, Vogelzang N, Stadler W, Hauke RJ, Monk JP, Saylor P, Bhoopalam N, Saad F, Sanford B, Kelly WK, Morris M, Small EJ. Randomized controlled trial of early zoledronic acid in men with castration-sensitive prostate cancer and bone metastases: results of CALGB 90202 (alliance). J Clin Oncol. 2014 Apr 10;32(11):1143-50. doi: 10.1200/JCO.2013.51.6500. Epub 2014 Mar 3. PMID 24590644
- [Result] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Result] Saad F, Shore N, Van Poppel H, Rathkopf DE, Smith MR, de Bono JS, Logothetis CJ, de Souza P, Fizazi K, Mulders PF, Mainwaring P, Hainsworth JD, Beer TM, North S, Fradet Y, Griffin TA, De Porre P, Londhe A, Kheoh T, Small EJ, Scher HI, Molina A, Ryan CJ. Impact of bone-targeted therapies in chemotherapy-naive metastatic castration-resistant prostate cancer patients treated with abiraterone acetate: post hoc analysis of study COU-AA-302. Eur Urol. 2015 Oct;68(4):570-7. doi: 10.1016/j.eururo.2015.04.032. Epub 2015 May 16. PMID 25985882
- [Result] Beer TM, Armstrong AJ, Rathkopf DE, Loriot Y, Sternberg CN, Higano CS, Iversen P, Bhattacharya S, Carles J, Chowdhury S, Davis ID, de Bono JS, Evans CP, Fizazi K, Joshua AM, Kim CS, Kimura G, Mainwaring P, Mansbach H, Miller K, Noonberg SB, Perabo F, Phung D, Saad F, Scher HI, Taplin ME, Venner PM, Tombal B; PREVAIL Investigators. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Jul 31;371(5):424-33. doi: 10.1056/NEJMoa1405095. Epub 2014 Jun 1. PMID 24881730
- [Result] Vanel D, Casadei R, Alberghini M, Razgallah M, Busacca M, Albisinni U. MR imaging of bone metastases and choice of sequence: spin echo, in-phase gradient echo, diffusion, and contrast medium. Semin Musculoskelet Radiol. 2009 Jun;13(2):97-103. doi: 10.1055/s-0029-1220880. Epub 2009 May 19. PMID 19455472
- [Result] Ma J. Dixon techniques for water and fat imaging. J Magn Reson Imaging. 2008 Sep;28(3):543-58. doi: 10.1002/jmri.21492. PMID 18777528
- [Result] Mosavi F, Johansson S, Sandberg DT, Turesson I, Sorensen J, Ahlstrom H. Whole-body diffusion-weighted MRI compared with (18)F-NaF PET/CT for detection of bone metastases in patients with high-risk prostate carcinoma. AJR Am J Roentgenol. 2012 Nov;199(5):1114-20. doi: 10.2214/AJR.11.8351. PMID 23096187
- [Result] Padhani AR, Makris A, Gall P, Collins DJ, Tunariu N, de Bono JS. Therapy monitoring of skeletal metastases with whole-body diffusion MRI. J Magn Reson Imaging. 2014 May;39(5):1049-78. doi: 10.1002/jmri.24548. Epub 2014 Feb 10. PMID 24510426
- [Result] Huang W, Li X, Chen Y, Li X, Chang MC, Oborski MJ, Malyarenko DI, Muzi M, Jajamovich GH, Fedorov A, Tudorica A, Gupta SN, Laymon CM, Marro KI, Dyvorne HA, Miller JV, Barbodiak DP, Chenevert TL, Yankeelov TE, Mountz JM, Kinahan PE, Kikinis R, Taouli B, Fennessy F, Kalpathy-Cramer J. Variations of dynamic contrast-enhanced magnetic resonance imaging in evaluation of breast cancer therapy response: a multicenter data analysis challenge. Transl Oncol. 2014 Feb 1;7(1):153-66. doi: 10.1593/tlo.13838. eCollection 2014 Feb. PMID 24772219
- [Result] Malyarenko DI, Zimmermann EM, Adler J, Swanson SD. Magnetization transfer in lamellar liquid crystals. Magn Reson Med. 2014 Nov;72(5):1427-34. doi: 10.1002/mrm.25034. Epub 2013 Nov 20. PMID 24258798
- [Result] Tombal B, Borre M, Rathenborg P, Werbrouck P, Van Poppel H, Heidenreich A, Iversen P, Braeckman J, Heracek J, Baskin-Bey E, Ouatas T, Perabo F, Phung D, Baron B, Hirmand M, Smith MR. Long-term Efficacy and Safety of Enzalutamide Monotherapy in Hormone-naive Prostate Cancer: 1- and 2-Year Open-label Follow-up Results. Eur Urol. 2015 Nov;68(5):787-94. doi: 10.1016/j.eururo.2015.01.027. Epub 2015 Feb 14. PMID 25687533